CLINICAL TRIAL: NCT01947569
Title: Autologous Co-stimulation-impaired Dendritic Cells for Type 1 Diabetes Mellitus (T1DM) Therapy: A Sequential Open Label Phase IB Safety Assessment/ Randomized, Double-blind Phase IIA Efficacy Trial to Maintain and Improve Functional Beta Cell Mass in New Onset Disease T1DM Patients
Brief Title: Dendritic Cells for Type 1 Diabetes Mellitus (T1DM) Therapy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: DiaVacs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DV-0100-100
Record Dates: First submitted 2013-09-18; First posted 2013-09-20 (Estimated); Last update posted 2013-10-23 (Estimated); Status verified 2013-10

CONDITIONS: Treatment of Type I Diabetes Mellitus.
MeSH Terms: interventions — Biological Products

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- iDC recipients (Experimental): iDC cells modified by in vitro engineering.
  Interventions: Biological: Biological
- Control DC recipients (Active Comparator): DC cells which have not been modified.
  Interventions: Biological: Biological
- Placebo recipients (Placebo Comparator): Saline injections.
  Interventions: Biological: Biological

INTERVENTIONS:
Biological: Biological

SUMMARY:
Phase IB will evaluate the safety of autologous, ex vivo-engineered, co-stimulation impaired dendtritic cells to maintain and improve functional residual beta cell mass in new onset Type I Diabetes Mellitus (T1DM) patients. Efficacy measures will be collected and summarized.

Phase IIA will evaluate the safety and efficacy of 3 randomized treatment groups in new onset T1DM patients to assess if the antisense DNA-treated co-stimulation-impaired immunoregulatory dendritic cells (iDC) will safely preserve and/or increase B-cell mass resulting in improvement and/or normalization of blood glucose levels and glycated hemoglobin A1c.

ELIGIBILITY:
Inclusion Criteria:(both open label phase IB safety and Phase IIA study):

1. Patients with new onset T1DM (>18 years of age for the phase IB and then >16 (first 10 subjects), >12 years of age for the second 10 subjects, > 8 years for the next 10 subjects and, finally, >8 years of age for the remainder of the phase IIA patients) within 6 months of diabetes mellitus diagnosis.
2. Evidence of decreased β-cell function as measured by C-peptide and blood glucose levels consistent with impaired glucose tolerance.
3. Evidence of at least one high-risk HLA haplotype.
4. Evidence of at least one diabetes-related autoantibody (e.g. IA-2, GAD, ZnT8) ,
5. Adequate immune competence as assessed by immunoreactivity to alloantigens in mixed leukocyte culture and reactivity to viral antigens (CEF Pool Assay) in vitro.
6. Normal hematologic, liver and kidney function.
7. Female participants of childbearing potential in this study must agree to use an effective form of birth control during study participation. Reliable and effective forms of birth control include: true abstinence, intrauterine device (IUD), hormonal-based contraception, double-barrier contraception [condom or occlusive cap (diaphragm or cervical cap) with spermicide], or surgical sterilization (vasectomy for male partner, tubal ligation or hysterectomy). Sexually active male participants must agree to use an effective form of birth control such as condoms.

Exclusion Criteria:(both open label phase IB safety and Phase IIA study):

1. Enrollment or history of enrollment in a drug, or biologic therapy study sponsored by TrialNet.
2. A significant history or current evidence of cardiac disease, uncontrolled hypertension, serious arrhythmias.
3. Evidence of active infection requiring antibiotic therapy.
4. History of other concurrent significant medical diseases.
5. Pregnant or lactating women.
6. Patients requiring chronic systemic corticosteroids.
7. Any other immune disorder including but not limited to other autoimmune diseases, HIV, HBV, HCV, HPV, HSV positivity.
8. Impaired renal function with a creatinine level > 1.5.
9. Administration of the following therapies while patients are undergoing treatment on this protocol: i) radiation therapy; ii) chemotherapy; iii) corticosteroids (except when administered in life-threatening circumstances); iv) other particle or cell-based therapies; v) other biologic therapies; vi) other therapies aimed at modulating the immune system; vii) other endocrine-related therapies, hormone replacement (other than thyroxine and contraceptive), glucoregulation.
10. A hemaglobinopathy known to interfere with the ability to accurately determine HbA1c.
11. No prior radiation therapy, immunotherapy, or chemotherapy.

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
The incidence of treatment-emergent adverse events. | Month 12

SECONDARY OUTCOMES:
2-hour area under the curve (AUC) average of C-peptide at 12 months after completion of administration of assigned therapy (Protocol Month 15). | 12 Months

CONTACTS AND LOCATIONS:
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States